CLINICAL TRIAL: NCT01371695
Title: Phase 1 of Serum IGF II and Cancer: Can IGF II Levels be Used to Monitor and Screen Patients Specifically for Cervical Cancer
Brief Title: Serum IGF-II and Cancer: Can IGF II Levels be Used to Monitor and Screen Patients Specifically for Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Onconix, Inc (Industry)
Responsible Party: Sharad A. Ghamande, Georgia Health Sciences University
Other Study IDs: onc11-03-164
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2011-06

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia II; Cervical Intraepithelial Neoplasia III
Keywords: IGF-II levels
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — frozen serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether Insulin-like Growth Factor II is elevated sufficiently to detect Cervical Intraepithelial Neoplasia II (CIN II), Cervical Intraepithelial Neoplasia III (CIN III), and cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years
* Female
* Normal medical history
* Medical history of a single type of cancer confirmed by biopsy or equivalent criteria
* Squamous cell carcinoma of organs other than cervix
* Adenocarcinoma
* Medical history of inflammatory disease
* May be pregnant
* Pap smear positive for Cervical Intraepithelial Neoplasia II or III
* Squamous cell cervical cancer confirmed by biopsy
* Informed consent
* Willingness to submit a blood sample by venipuncture
* Willingness to submit a second blood sample if necessary

Exclusion Criteria:

* Age < 18 or > 75 years
* Medical history of cancer other than cervical cancer, Non-islet-cell tumor hypoglycemia, Growth hormone deficiency, Acromegaly, Hepatoma, inflammatory disease in addition to confirmed CIN and cervical cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: university clinic
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Estimated); Study Completion 2013-09 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Georgia Health Sciences, Augusta, Georgia, United States